CLINICAL TRIAL: NCT02937623
Title: A Proof-of-principle Clinical Study Investigating the Efficacy of a Dissolvable Strip in Providing Rapid Relief From Dentinal Hypersensitivity.
Brief Title: To Evaluate the Efficacy of an Experimental Dissolvable Strip in Rapidly Relieving Dentinal Hypersensitivity (DH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 207238
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Test Product: Dissolvable polymer strip containing Novamin (Experimental): In this arm, participants received an experimental dissolvable polymer strip containing 15 % weight/weight (w/w) calcium sodium phosphosilicate (Novamin). One strip was applied per test tooth topically by a suitably qualified member of the site staff. Each participant received 2 strips in total (as two test tooth were assessed per participant).
  Interventions: Device: Dissolvable polymer strip containing Novamin (calcium sodium phosphosilicate)
- Reference Product: No treatment/product (No Intervention): In this arm, participants did not receive any treatment/product.

INTERVENTIONS:
Device: Dissolvable polymer strip containing Novamin (calcium sodium phosphosilicate) — Experimental dissolvable polymer strip containing Novamin (15% weight by weight[w/w] calcium sodium phosphosilicate).
  Arms: Test Product: Dissolvable polymer strip containing Novamin

SUMMARY:
A proof of principle single-centre, randomized-controlled, examiner-blind, two treatment group study to investigate the efficacy of an experimental 15% w/w dissolvable strip in relieving dentine hypersensitivity (DH) after a single application and up to 4 hours after application compared to no treatment.

DETAILED DESCRIPTION:
This was a single-centre, randomized-controlled, examiner-blind, two treatment group (test and no treatment), parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected test teeth) study, in healthy participants with at least two sensitive teeth that meet all the criteria at the screening and the baseline pre-treatment visit. Participants were screened for study suitability at screening visit (Visit 1). At Visit 2 (baseline; pre-treatment) 2 non-adjacent accessible teeth (incisors, canines, premolars) in different quadrants of the mouth and separated by at least 2 teeth (or equivalent edentulous space) were identified that demonstrated signs of sensitivity as measured by a qualifying tactile stimulus (Yeaple ≤ 20 gram [g]) and evaporative air assessment (Schiff sensitivity score ≥ 2) on the facial/cervical (ie, labial/buccal) tooth surface. Once the 2 test teeth were selected, the subjects were stratified (by maximum baseline Schiff sensitivity score of the 2 selected test teeth) and randomized to treatment or no treatment. DH was assessed at baseline (pre-treatment), and 10mins, 2 & 4 hours post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received assigned and dated copy of the informed consent form.
* Aged 18-65 years.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities of medical history or oral Examination and absence of any condition that would impact on the participants safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* At Visit 1 (Screening): a) Self-reported history of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years. b) Minimum of 20 natural teeth. c) Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), in different quadrants and separated by at least two teeth (or equivalent edentulous space), that meet all of the following criteria: Signs of facial/ cervical (i.e. labial/ buccal) gingival recession and/or signs of erosion or abrasion (EAR), tooth with MGI score = 0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1 and tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response) on the facial/ cervical (i.e. labial/ buccal) tooth surface.
* At Visit 2, Baseline (Pre-treatment): Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars) in different quadrants of the mouth and separated by at least two teeth (or equivalent edentulous space), that meet all of the following criteria: Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff sensitivity score ≥ 2) on the facial/ cervical (i.e. labial/ buccal) tooth surface.

Exclusion Criteria:

* A woman who is known to be pregnant or who are intending to become pregnant over the duration of the study.
* A women who is breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit and previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes and any condition which, in the opinion of the investigator, causes xerostomia (dry mouth).
* Dental prophylaxis within 4 weeks of Screening, tongue or lip piercing, desensitizing treatment within 8 weeks of Screening (professional sensitivity treatments and non-dentifrice sensitivity treatments), gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of screening, scaling or root planning within 3 months of screening and teeth bleaching within 8 weeks of screening.
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of screening and tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, dental implants, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine. Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening (Participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients).
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs, currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline and daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Gallob J, Ling MR, Amini P, Patil A, Atassi M. Efficacy of a dissolvable strip with calcium sodium phosphosilicate (NovaMin(R)) in providing rapid dentine hypersensitivity relief. J Dent. 2019;91S:100003. doi: 10.1016/j.jjodo.2019.100003. Epub 2019 Jun 15. PMID 34059276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in USA.
Pre-assignment Details: A total of 135 participants were screened, out of which 126 were enrolled in study. 9 participants were screening failure so did not enrolled. Out of 126 enrolled participants, 120 participants were randomized. 6 participants were not randomized as 1 had adverse event, 3 withdrew from study before randomization & 2 because of unspecified reasons.
Period: Overall Study
Arm/Group | Test Product: Dissolvable Polymer Strip Containing Novamin | Reference Product: No Treatment/Product
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test Product: Dissolvable Polymer Strip Containing Novamin: In this arm, participants received an experimental dissolvable polymer strip containing 15 % w/w calcium sodium phosphosilicate (Novamin). One strip was applied per test tooth topically by a suitably qualified member of the site staff. Each participant received 2 strips in total (as two test tooth were assessed per participant).
- Total: Total of all reporting groups
Arm/Group | Test Product: Dissolvable Polymer Strip Containing Novamin | Reference Product: No Treatment/Product | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.75) | 38.8 (11.36) | 38.2 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 20 | 21 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 15 | 25 | 40
  White | 34 | 26 | 60
  More than one race | 4 | 8 | 12
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score After 10 Minutes
Description: The examiner indicated the participant's response to the evaporative air stimulus, after the stimulation of each test tooth, using the Schiff Sensitivity Scale as follows: 0= Participant does not respond to air stimulation, 1= Participant responds to air stimulus but does not request discontinuation of stimulus, 2= Participant responds to air stimulus and requests discontinuation or moves from stimulus, 3= Participant responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicate improvement in sensitivity.
Time Frame: At baseline (pre-treatment) and 10 minutes post-treatment: Day 1 of the study
Population: Intent-to-treat (ITT) population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product: Dissolvable Polymer Strip Containing Novamin | Reference Product: No Treatment/Product
Number analyzed (Participants) | 60 | 60
score on a scale | -0.46 (0.531) | -0.02 (0.260)
Statistical Analysis 1: Comparison: Test Product: Dissolvable Polymer Strip Containing Novamin vs Reference Product: No Treatment/Product; Test type: Other; p < .0001, ANCOVA; ANCOVA model: change from baseline in Schiff sensitivity score as response and treatment as factors and baseline Schiff sensitivity score as covariate; Least square mean difference = -0.44, 95% CI [-0.591 to -0.297] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favours first named dentifrice

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score After 2 and 4 Hours
Description: as for outcome 1
Time Frame: At Baseline (pre-treatment), 2 and 4 hours post-treatment: Day 1 of the study
Population: ITT population included all participants who were randomized, received the study treatment at least once and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product: Dissolvable Polymer Strip Containing Novamin | Reference Product: No Treatment/Product
Number analyzed (Participants) | 60 | 60
score on a scale
  Change from baseline after 2 hours | -0.78 (0.654) | -0.08 (0.334)
  Change from baseline after 4 hours | -1.03 (0.698) | -0.12 (0.361)

3. Secondary Outcome: Change From Baseline in Tactile Threshold After 10 Minutes, 2 Hours and 4 Hours
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force has reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline (pre-treatment), the maximum force used was 20g; at all subsequent time points (post treatment), it was 80g.
Time Frame: At Baseline (pre-treatment), 10 minutes, 2 hours and 4 hours post treatment: Day 1 of the study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Test Product: Dissolvable Polymer Strip Containing Novamin | Reference Product: No Treatment/Product
Number analyzed (Participants) | 60 | 60
gram (g)
  Change from baseline after 10 minutes | 8.92 (10.580) | 0.50 (2.383)
  Change from baseline after 2 hours | 16.50 (16.424) | 0.75 (2.405)
  Change from baseline after 4 hours | 24.00 (20.704) | 0.92 (2.346)

4. Secondary Outcome: Change From Baseline in Numerical Rating Scale (NRS) Scores After 10 Minutes, 2 Hours and 4 Hours
Description: Participants rated the intensity of their response to the evaporative air stimulus using a 10 point numerical rating scale of 1 (No Pain) to 10 (Intense Pain).
Time Frame: At baseline(pre-treatment), 10 minutes, 2 hours and 4 hours post treatment: Day 1 of the study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Test Product: Dissolvable Polymer Strip Containing Novamin | Reference Product: No Treatment/Product
Number analyzed (Participants) | 60 | 60
score on a scale
  Change from baseline after 10 minutes | -1.44 (1.571) | -0.11 (0.893)
  Change from baseline after 2 hours | -1.92 (1.762) | -0.47 (1.149)
  Change from baseline after 4 hours | -2.49 (1.917) | -0.33 (0.896)

ADVERSE EVENTS:
Arm/Group | Test Product: Dissolvable Polymer Strip Containing Novamin | Reference Product: No Treatment/Product
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.